CLINICAL TRIAL: NCT01388595
Title: A Proof of Concept Study to Evaluate Effects of Intranasal Salmeterol and Fluticasone Given Alone and in Combination in Allergic Rhinitis
Brief Title: Fluticasone and Salmeterol in Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NAI002
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Therapeutics; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fluticasone Proprionate (Active Comparator): The participants will be randomised and at each study visit, will receive a single inhaler which can either be active or placebo.
  Interventions: Drug: FLUTICASONE PROPRIONATE
- Salmeterol (Active Comparator): The participants will be randomised and at each study visit, will receive a single inhaler which can either be active or placebo.
  Interventions: Drug: Salmeterol
- placebo (Placebo Comparator): The participants will be randomised and at each study visit, will receive a single inhaler which can either be active or placebo.
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: FLUTICASONE PROPRIONATE — 1. Fluticasone Propionate (FP) Product name: Flixotide Evohaler® Manufacturer: Allan and Hanbury's Active ingredients: Fluticasone Propionate Propellant: HFA 134a Dose: 250μg per actuation giving a total dose of 500µg per day through the spacer device with the customised nasal adaptor.
  Other Names: Treatment
  Arms: Fluticasone Proprionate
Drug: Salmeterol — Salmeterol Product Name: Serevent® Manufacturer: Allan and Hanbury's Active ingredients: Salmetrol Xinafoate Propellant: HFA 134a Dose: 25μg per actuation giving a total dose of 50µg per day through the spacer device with the customised nasal adaptor
  Other Names: Treatment
  Arms: Salmeterol
Drug: PLACEBO — 4. Placebo inhaler to SM, FP, SM+FP Manufacturer: Cipla Ltd Active ingredients: None Propellants: HFA 134a Imported & QP release tested in UK : DHP Clinical supplies, Powys, UK
  Other Names: Treatment
  Arms: placebo

SUMMARY:
Allergic rhinitis is an under diagnosed global health problem which affects up to 25% of the population worldwide. It has been reported as being one of the 10 most common causes for attendance to primary care clinics. It is clinically defined as a symptomatic disorder of the nose induced by an IgE mediated inflammation following allergen exposure of the membranes lining the nose and is characterized by varying combinations of nasal symptoms including sneezing, nasal blockage, rhinorrhoea and itching. Intra nasal corticosteroids form the cornerstone of anti-inflammatory therapy in allergic rhinitis and there is increasing interest in the role of intranasal beta 2 agonists in the management of allergic rhinitis. The question therefore arises as to whether salmeterol exhibits such synergistic activity in the nose in terms of potentiating the steroid response of fluticasone.

DETAILED DESCRIPTION:
In vitro and ex vitro data have suggested that salmeterol may exhibit ligand independent activation of glucocorticoid receptors, which might result in potentiation of fluticasone by salmeterol when given in combination.

Although no such evidence of synergy was reported with fluticasone salmeterol combination in the nose with allergen challenge, no data are available on nasal AMP challenge in the nose.

This study compares the single and long term dosing effects of intranasal fluticasone alone, salmeterol alone and fluticasone salmeterol combination on nasal AMP challenge in persistent allergic rhinitis sufferers.

Nasal corticosteroid,leukotriene receptor antagonist and anti histamine stopped for one week before the start of randomized treatment during the run in phase and wash out periods. Intransal sodium cromoglycate spray provided for rescue use throughout the study but witheld for at least twenty four hours before challenge.

Nasal AMP challenges performed at baseline, after run-in and each washout, and 12 hours after the first and last evening dose of the study medication. A Zerostat Antistatic spacer (Cipla, Mumbai, India) used to administer the randomized treatments, adapted with a nasal olive for intranasal use instead of the conventional mouthpiece.

The randomized treatments given once daily at night time as follows: placebo hydrofluoroalkane, 2 puffs (Cipla, Mumbai,India) salmeterol-hydrofluoroalkane, 2 puffs of 25 g (Serevent Evohaler Allen and Hanburys, Middlesex, United Kingdom) fluticasone- salmeterol hydrofluoroalkane, 2 puffs of 250/25 g (Seretide Evohaler, Allen and Hanburys) and fluticasone-hydrofluoroalkane,2 puffs of 250 g (Flixotide Evohaler, Allen and Hanburys).

The double-blind randomization process computer generated from www.randomization.com. Trial drug randomization performed under the direct supervision of the clinical trial pharmacist at Ninewells University Hospital.

Active fluticasone,salmeterol, and fluticasone-salmeterol combination procured from GlaxoSmithKline (Allen and Hanburys) by the clinical trial pharmacy and matched placebo provided by Cipla.

Following Informed Consent and screening visit, participants provided with randomized, labeled treatment packs with a single inhaler, either active or placebo at each study treatment visit.

Blinding of patients and investigators ensured by using identical colored actuators for each treatment and labeling of active or placebo canisters with trial-specific labels.

Measurements made at 12 hours after the first and last dose of each randomized treatment.

At initial screening, nasal endoscopy performed to exclude significant nasal polyp disease (greater than grade 1), concha bullosa, and septal deviation.

A Niox Flex nitric oxide analyzer (Aerocrine AB, Solna, Sweden) used to measure nasal nitric oxide. The standard aspiration technique recommended by the American Thoracic Society/European Respiratory Society guidelines used with a unilateral,nasal olive, breath-holding, and velum closure.

For nasal AMP challenge, PNIF measured before and every 5 minutes for 60 minutes after 4 squirts of 0.1 mL per actuation in each nostril of 400 mg/mL of AMP (ie, 320-mg total dose) delivered to the nose. The maximum decrease in PNIF measured using an In-check Nasal Inspiratory Flow Meter (Clement Clarke International Ltd, Harlow, United Kingdom).

It has been shown that measuring PNIF (PEAK NASAL INSPIRATORY FLOW) response is more sensitive than measuring nasal airway resistance and is also more reproducible.PNIF correlates well vs symptoms in response to treatment in allergic rhinitis patients and has been shown to have a minimal clinically important difference of 5 L/min.

At screening, patients instructed in the correct technique with particular attention to horizontal positioning of the meter, a closed mouth with maximal peak nasal inspiratory effort, and an adequate mask seal around the mouth and nose.

Nasal impulse oscillometry measurements for nasal airway resistance at 5 Hz performed using a Jaeger MasterScreen impulse oscillometry system (Erich Jaeger, Hoechberg, Germany).

The total nasal symptom 4 (TNS4) scores recorded at all visits, with a total score of 12 for the sum of the 4 separate domains for nasal blockage, run, itch, and sneeze, each rated from 0 to 3.

The Juniper Mini Rhinoconjunctivitis Quality of Life Questionnaire (Mini-RQLQ) completed by the participant immediately before and a week after each randomized treatment. The global RQLQ is the mean of the 5 individual domains, with individual domains scored from 0 to 6.

Serum eosinophilic cationic protein measured using an enzyme-linked immunoassay technique (UniCAP; Sweden Diagnostics UK Ltd, Milton Keyes, United Kingdom).

ELIGIBILITY:
Inclusion Criteria:

1. Persistent allergic rhinitis without asthma.
2. Atopy to at least 1 allergen on SPT.
3. ≥ 20% drop in PNIF following nasal AMP challenge
4. Male to female aged 18-65
5. Informed Consent
6. Ability to comply with the protocol

Exclusion Criteria:

1. Severe allergic rhinitis as defined by those in whom there are symptoms which significantly impair day to day activities on QOL questionnaire.
2. Nasal Polyposis grade 2/3, deviated nasal septum ≥ 50%
3. PNIF < 60 litres/min
4. The use of oral corticosteroids within the last 3 months.
5. Recent respiratory tract / sinus infection (2 months).
6. Significant concomitant respiratory disease such as COPD, CF, ABPA, bronchiectasis and active pulmonary tuberculosis.
7. Any other clinically significant medical condition such as unstable angina, acute myocardial infarction in the preceding 3 months, recent TIA/ CVA,that may endanger the health or safety of the participant, or jeopardise the protocol.
8. Any significant abnormal laboratory result as deemed by the investigators
9. Pregnancy, planned pregnancy or lactation
10. Known or suspected contra-indication to any of the IMP's
11. Concomitant use of medicines (prescribed, over the counter or herbal) that may interfere with the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in Peak Nasal Inspiratory Flow (PNIF). | Change from baseline at 1 week.
  Maximum change in PNIF following nasal adenosine monophoshate (AMP) challenge testing for active groups versus placebo.. Data will be presented as % change between groups.

SECONDARY OUTCOMES:
Nasal symptom scores. | Change from baseline at 1 week.
  Nasal Quality of Life Scoring.
Nasal nitric oxide. | Change from baseline at 1 week.
Nasal impulse oscillometry. | Change from baseline at 1 week.
  Assessment of airway resistance.
Eosinophil cationic protein (ECP) | Change from baseline at 1 week.
  Serum blood test
Overnight urinary cortisol/creatinine. | Change from baseline at 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Lipworth, MD, Principal Investigator — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, University of Dundee, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lipworth BJ, Short P, Burns P, Nair A. Effects of intranasal salmeterol and fluticasone given alone and in combination in persistent allergic rhinitis. Ann Allergy Asthma Immunol. 2012 Jan;108(1):54-59. doi: 10.1016/j.anai.2011.10.001. Epub 2011 Nov 2. PMID 22192967